CLINICAL TRIAL: NCT05273814
Title: Phase I Clinical Study of Tislelizumab in Combination With Bevacizumab and Pemetrexed for the First-line Treatment of Advanced Non-squamous Non-small Cell Lung Cancer in Elderly Patients
Brief Title: Study of Chemotherapy and PD-1 Inhibitor Combination With Anti-angiogenesis to Treat Elderly Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCICC-005
Record Dates: First submitted 2022-01-28; First posted 2022-03-10 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Immune Checkpoint Inhibitors; Pemetrexed; Drug Therapy; Bevacizumab; Angiogenesis Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab+Bevacizumab+Pemetrexed (Experimental): Bevacizumab，7.5mg/kg，d1; Pemetrexed，500mg/m2，d1; Tislelizumab，200mg，d4; Q3W for 4 cycles;
  Maintenance treatment ： Tislelizumab，200mg，d1; Bevacizumab，7.5mg/kg，d1; Q3W for 2 years
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed; Drug: Bevacizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab intravenous infusion 200mg d4
  Other Names: PD-1 inhibitor
Drug: Pemetrexed — Pemetrexed intravenous infusion 500mg/m2 d1
  Other Names: Chemotherapy
Drug: Bevacizumab — Pemetrexed intravenous infusion 7.5mg/kg，d1
  Other Names: Anti-angiogenesis

SUMMARY:
This single-center, open-label, phaseⅠstudy is to evaluate the efficacy of Tislelizumab in combination with Bevacizumab and Pemetrexed for the first-line treatment of advanced Non-squamous Non-small Cell lung cancer in Elderly Patients

DETAILED DESCRIPTION:
Patients received Bevacizumab, 7.5mg/kg d1, Pemetrexed, 500mg/m2, d1 and Tislelizumab 200mg, d4, Q3W, for 4 cycles; then Tislelizumab 200mg, d1 Q3w and Bevacizumab 7.5mg/kg d1 Q3W, maintenance treatment for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Subjects who must meet all the following criteria should be selected:

1. Agree to participate in this trial and sign written informed consent form.
2. Male or female, age ≥ 65 years.
3. Expected survival time ≥ 3 months and able to be followed-up.
4. Stage IIIB/IIIC/IV non-squamous NSCLC patients without previous systemic therapy (according to AJCC8th) or patients with stage IIIB/IIIC/IV non-squamous NSCLC who have relapsed after surgery (if adjuvant therapy was administered, more than 6 months of drug discontinuation is required).
5. Without EGFR mutation and ALK and ROS1 fusion genes.
6. Patients can not receive concurrent chemoradiothrapy after multidisciplinary consultation and discussion.
7. At least one measurable tumor indicator along with a lesion with a maximum diameter of ≥ 1 cm (diagnosed by imaging, e.g., CT, MRI, ECT).
8. ECOG PS 0-1 within 7 days before enrollment.
9. Within 14 days prior to the start of treatment, laboratory results of routine blood, liver and kidney function and hormone levels meet the following criteria: platelets (PLT) ≥ 100 × 109/L, neutrophils (ANC) ≥ 1.5 × 109/L, hemoglobin (HGB) ≥ 90 g/L, aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN) (≤ 5 × ULN for liver metastases), alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for liver metastases), total bilirubin (TIBC) ≤ 1.5 × ULN, and alanine aminotransferase (ALT) ≤ 1.5 × ULN. × ULN), alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for liver metastases), total bilirubin (TIBC) ≤ 1.5 × ULN, serum creatinine (CR) ≤ 1.25 × ULN; cortisol and thyroid function are in the normal range.
10. Toxic effects of prior chemotherapy have resolved to grade 1 or less (except alopecia). Subjects must have recovered from toxicity or complications of these interventions if they have received major surgical treatment or > 30Gy of radiation therapy, i.e., they are still eligible for enrollment after 6 months.

Exclusion Criteria:

Subjects who meet any of the following criteria could not participate in this study:

1. Received bevacizumab and/or pemetrexed within 6 months prior to the first dose of study drug.
2. Other malignant tumors with disease progression or requiring aggressive treatment within 5 years of enrollment. Exceptions included early-stage tumors (carcinoma in situ or stage I tumors) that received radical treatment, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the breast that received potentially radical treatment.
3. Have had an allogeneic tissue/organ transplant.
4. Participating or have participated in investigational drug therapy within 4 weeks prior to the first dose of the trial.
5. Receiving systemic hormone therapy or are receiving any other form of immunosuppressive therapy (except docetaxel pretreated glucocorticoids) within 14 days prior to the first dose of the experimental treatment.
6. Received anti-tumor monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or major surgical procedure within 1 month prior to the first use of study drug; received chest radiation therapy greater than 30 Gy within 6 months prior to the first use of study drug; received chest radiation therapy at 30 Gy or less within 1 month prior to the first use of study drug.
7. Prior treatment with other PD-1 antibodies and other immunotherapy targeting PD-1/PD-L1.
8. Active autoimmune disease requiring systemic therapy (e.g., use of disease-relieving drugs, corticosteroids, or immunosuppressants) within the past 2 years Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic therapy.
9. Having congenital or acquired immune deficiency (e.g., HIV-infected patients), active hepatitis B (HBV-DNA ≥ 2.5 x 10^3 copies/ml), or hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of detection for the assay).
10. Patients who have received live vaccine within 4 weeks prior to the first administration of study drug are permitted to receive inactivated viral vaccine for seasonal influenza, administered by injection, but not live attenuated influenza vaccine administered via the nose.
11. Patients with known active central nervous system (CNS) metastases and/or cancerous meningitis. Subjects who have had treatment for brain metastases may also participate in this study provided that the subject is stable (no evidence of progression for at least 4 weeks and all neurological symptoms have returned to baseline levels as determined by MRI prior to the first dose), has no evidence of new or expanding brain metastases, and has not used hormone therapy for at least 3 days prior to study dosing.
12. Bleeding tendency, high bleeding risk, or coagulopathy with a history of thrombotic disease within 6 months and/or hemoptysis within 3 months; being treated with full doses of oral and/or parenteral anticoagulants and thrombolytics (prophylactic anticoagulation is allowed); having used aspirin or other non-steroidal anti-inflammatory drugs that inhibit platelet function within 10 days; and CT/MRI imaging showing tumor encapsulation or invasion of the lumen of large blood vessels.
13. Poorly controlled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg) and patients with prior hypertensive crisis and hypertensive encephalopathy; severe cerebrovascular disease.
14. Non-healing wounds, peptic ulcers in active phase, tracheo-esophageal fistulas, gastrointestinal perforations and intra-abdominal abscesses within 6 months.
15. Have an active infection that requires systemic treatment via Intravenous injection.
16. Have mental illness or other condition, such as uncontrolled heart or lung disease, diabetes mellitus, etc., that prevents cooperation with study treatment and monitoring requirements.
17. History of interstitial lung disease.
18. Patients with moderate to heavy smoking need to quit smoking for more than 1 month.
19. Known allergy to any of the components of the study drug.
20. Patients who are regular users of any drug (including "recreational" use) or have recent history (within 1 year) of substance abuse (including alcohol) when signing the informed consent form.
21. Poor compliance and inability to cooperate with the clinical study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | approximately 2 years
  ORR was calculated by the percentage of patients with a confirmed complete (CR) or partial response (PR).

SECONDARY OUTCOMES:
Overall survival | approximately 3 years
  Time from the first use of the study drug to the death of the subject
Progression-free survival | approximately 2 years
  Progression-free survival is defined as the time from the start of treatment to the first documentation of disease progression or death from any cause, whichever occurs first according to RECIST 1.1.
Duration of response | approximately 2 years
  Duration of response is defined as the time from the first recording of evidence of CR or PR until disease progression (according to RECIST 1.1) or death from any cause, whichever occurs first
Health-related quality of life | approximately 2 years
  Measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer Core 30 (EORTC QLQ-C30) as presented in participants-reported outcomes.Scale construct including to assess Global health status/QoL with range from minimum scores 1 as worse outcome and maximum scores 7 as higher values represent a better; Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning, Fatigue, Nausea and vomiting, Pain Dyspnoea, Insomnia, Appetite loss, Constipation, Diarrhoea and Financial difficulties with range from maximum scores 4 as worse outcome and from minimum scores 1 as higher values represent a better.
Safety and tolerance | approximately 2 years
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol